CLINICAL TRIAL: NCT03611218
Title: Comparative Safety and Clinical Performance of Dialyzers Applied During Post-dilution Online Hemodiafiltration - eMPORA II Study (Modified POlysulfone membRAne)
Brief Title: Comparative Safety and Clinical Performance of Dialyzers Applied During Post-dilution Online Hemodiafiltration
Acronym: eMPORA II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fresenius Medical Care Deutschland GmbH (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HD-FX-06-D
Record Dates: First submitted 2018-07-27; First posted 2018-08-02 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Renal Failure; End Stage Renal Disease
Keywords: Hemodialysis; Hemodiafiltration; Renal replacement therapy
MeSH Terms: conditions — Renal Insufficiency; Kidney Failure, Chronic | interventions — Kidneys, Artificial

STUDY DESIGN:
Intervention Model Description: Prospective, open, controlled, cross-over (with randomized treatment sequences), interventional, multi-center
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hemodiafiltration HDF (Other): Three consecutive treatment weeks and on follow-up week per patient. Each treatment week includes three hemodiafiltration HDFsessions and is assigned to one type of dialyzer: FX P600 Fresenius Medical Care, comparator Nipro: Sureflux-17UX and comparator Baxter/Gambro: Polyflux 170 H.
  Interventions: Device: Dialyzer

INTERVENTIONS:
Device: Dialyzer — Three hemodiafiltration sessions assigned to one type of dialyzer FX P600 (Fresenius Medical Care), comparator Sureflux-17UX and comparator Polyflux 170 H

SUMMARY:
The clinical Investigation will be performed to compare the safety and clinical performance profile of different hemodialyzers, all applied in on-line postdilution hemodiafiltration

DETAILED DESCRIPTION:
The primary objective of this study is to test whether the new FX P600 (applied during post-dilution online HDF) is non-inferior to two comparator dialyzers (Sureflux-17UX (Nipro) and Polyflux 170 H (Baxter/Gambro) in removing β2-microglobulin. The secondary objective is to exploratively compare the efficacy in removing other uremic solutes between the new FX P600 and the Sureflux-17UX as well as the Polyflux 170 H membranes. Additionally, the safety of the FX P600 dialyzer with a modified polysulfone membrane will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years
* Existing informed consent form signed and dated by study patient as well as investigator/authorized physician
* The patient is legally competent and able to understand the nature, risks, meaning, and consequences of the clinical trial and can subsequently declare his consent for participation in the clinical trial
* Patients with a chronic kidney disease stage 5D (end stage renal disease with a glomerular filtration rate of 15 ml/min or less) on hemodiafiltration as extracorporeal renal replacement therapy

Exclusion Criteria:

* Any condition which could interfere with the patient's ability to comply with the study. This decision is at the discretion of the treating physician and relates to the general stable condition of the patient (e.g. absence of any acute condition, e.g. infection or mental problem which might give reason for concern etc.).
* Ongoing participation in an interventional clinical study during the preceding 30 days
* Previous participation in this study
* Pregnancy (pregnancy test will be conducted with female patients aged ≤ 55 years) or lactation period
* Patient is not able to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2018-12-08 (Actual); Study Completion 2018-12-08 (Actual)

PRIMARY OUTCOMES:
Removal rate of β2-microglobulin | t=240 minutes of HDF
  Removal rate of β2-microglobulin will be calculated as primary endpoint in blood samples to evaluate the clinical performance of the new FX P600 dialyzer.

SECONDARY OUTCOMES:
Clearance of β2-microglobulin | t=60 minutes of HDF
Removal rate of α1-microglobulin | t=240 minutes of HDF
Clearance of α1-microglobulin | t= 60 minutes of HDF

CONTACTS AND LOCATIONS:
Locations (6):
- Germany (6):
  - Zentrum für Nieren-, Hochdruck- und Stoffwechselerkrankungen, Hanover, Lower Saxony
  - Diakonissenkrankenhaus Flensburg, Flensburg
  - Georg-Haas-Dialysezentrum der PHV, Giessen
  - PHV-Dialysezentrum Goslar, Goslar
  - PHV Dialysezentrum Kiel, Kiel
  - PHV-Dialysezentrum Lauterbach, Lauterbach

REFERENCES:
- [Derived] Ehlerding G, Erlenkotter A, Gauly A, Griesshaber B, Kennedy J, Rauber L, Ries W, Schmidt-Gurtler H, Stauss-Grabo M, Wagner S, Zawada AM, Zschatzsch S, Kempkes-Koch M. Performance and Hemocompatibility of a Novel Polysulfone Dialyzer: A Randomized Controlled Trial. Kidney360. 2021 Apr 7;2(6):937-947. doi: 10.34067/KID.0000302021. eCollection 2021 Jun 24. PMID 35373083